CLINICAL TRIAL: NCT02937415
Title: Breath Carbon Monoxide Measurement Predicts Oxidative Stress Which Cause of Deteriorations of Lung Functions in Waterpipe Smokers
Brief Title: Carbon Monoxide and Oxidative Stress in Waterpipe Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mukremin Er, Mukremin Er, MD., Ataturk Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AtaturkTRH
Record Dates: First submitted 2015-12-19; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Waterpipe Smoking; Oxidative Stress
Keywords: carbon monoxide; oxidative stress; waterpipe smoking; cigarette smoking; pulmonary function test
MeSH Terms: conditions — Water Pipe Smoking; Cigarette Smoking | interventions — Respiratory Physiological Phenomena; Oxidative Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Waterpipe smokers group (Experimental): Three waterpipe cafes located in Ankara were visited. 50 waterpipe smokers aged 18-40 years, enrolled in the study and created the working group. At the same time, there were also cigarette smokers among these people. Breath carbon monoxide, pulmonary function tests were performed both before and after smoking waterpipe and parameters of oxidative stress and antioxidant status were measured in blood samples after smoking waterpipe.
  Interventions: Procedure: Breath carbon monoxide; Procedure: Pulmonary function tests.; Procedure: Oxidative stress and antioxidant status.
- Control group (Active Comparator): The control group consisted of 50 people of the same age and sex, who had never smoked neither cigarette nor waterpipe. Breath carbon monoxide, pulmonary function tests were performed and parameters of oxidative stress were measured in blood samples.
  Interventions: Procedure: Breath carbon monoxide; Procedure: Pulmonary function tests.; Procedure: Oxidative stress and antioxidant status.

INTERVENTIONS:
Procedure: Breath carbon monoxide — Breath carbon monoxide measurement.
Procedure: Pulmonary function tests. — Measurement of lung functions by blowing through a tube which measures flow and volumes of participant's lungs.
  Other Names: Spirometry
Procedure: Oxidative stress and antioxidant status. — Measurement of parameters of oxidative stress and antioxidant status in blood samples.

SUMMARY:
Waterpipe is a tool for smoking tobacco, which is thought to be less harmful than cigarette. Unfortunately, there aren't adequate studies about its harms to health that are threatening the young generation all over the world today. The objective of this study was to show the carbon monoxide (CO) levels in waterpipe smokers' breaths, whether can be used or not to reflect the changes of oxidative stress for this reason to predict harmful effects on the pulmonary functions.

DETAILED DESCRIPTION:
Waterpipe or hookah uses a different kind of tobacco, which is available in most Balkan countries, Middle East and South Asia. Popularity of smoking waterpipe among European, Canadian, and American young people has shown a dramatic rise over the past decade. The growing popularity of waterpipe use among U.S. teens and adults is evidenced by media reports and the recent rapid proliferation of waterpipe establishments (bars, cafes, or restaurants) in large cities and near college campuses. Typical waterpipes have the following components; a bowl where the tobacco is placed and heated, usually with burning embers or charcoal, a vase or smoke chamber which is partially filled with water, a pipe or stem connecting the bowl to the vase by a tube that carries the smoke down into the water, and a hose with a mouthpiece through which the smoke is drawn from the vase. As the smoker inhales, the tobacco smoke is sucked down from the bowl and then bubbles up through the water into the air of the smoke chamber and then through the hose to the smoker. At the end of a smoking session, the dirty water is thrown away and the waterpipe vase is refilled for the next user. Although each smoking session generally lasts about 45 to 60 minutes, it can also continue for several hours.

There is a misconception about smoking waterpipe that it is less harmful than cigarettes, and that's why smoking waterpipe is dramatically increasing especially among young people. While the adverse effects of smoking cigarette are widely described, there are just a few investigations about waterpipe and its effects. This study was designed to investigate the effects of smoking waterpipe on pulmonary functions and oxidative stress parameters.

ELIGIBILITY:
Inclusion Criteria:

* Participants who haven't determined major health problems,
* between ages 18-40.

Exclusion Criteria:

* Participants who under age 18 and above 40,
* pregnant women,
* individuals who have major health problems

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Breath Carbon Monoxide Level | Up to 4 months
  Levels of CO in breath will be measured in either waterpipe smokers or control group.

SECONDARY OUTCOMES:
A spirometric Test; FEV1 (Forced Expiratory Volume in One Second) Measurement. | Up to 4 months
  FEV1 Will Be Measured To Evaluation of Deterioration Levels of Pulmonary Functions in Either Waterpipe Smokers or Control Group.
A spirometric Test; FVC (Forced Vital Capacity) Measurement. | Up to 4 months
  FVC Will Be Measured To Evaluation of Deterioration Levels of Pulmonary Functions in Either Waterpipe Smokers or Control Group.
A spirometric Test; FEV1/FVC (Forced Expiratory Volume in One Second/Forced Vital Capacity) Measurement. | Up to 4 months
  FEV1/FVC Will Be Measured To Evaluation of Deterioration Levels of Pulmonary Functions in Either Waterpipe Smokers or Control Group.
A spirometric Test; PEF (Peak Expiratory Flow) Measurement. | Up to 4 months
  PEF Will Be Measured To Evaluation of Deterioration Levels of Pulmonary Functions in Either Waterpipe Smokers or Control Group.
A spirometric Test; FEF25-75 (Forced Expiratory Flow in 25-75%) Measurement. | Up to 4 months
  FEF25-75 Will Be Measured To Evaluation of Deterioration Levels of Pulmonary Functions in Either Waterpipe Smokers or Control Group.
Plasma TAS (Total Anti-Oxydant Status) Measurement. | Up to 4 months
  To Assessment of Anti-Oxidant Status: TAS Levels in Plasma Will Be Measured in Either Waterpipe Smokers or Control Group.
Plasma TOS (Total Oxydative Stress) Measurement. | Up to 4 months
  To Assessment of Oxidative Stress: TOS Levels in Plasma Will Be Measured in Either Waterpipe Smokers or Control Group.
Plasma OSI Measurement. | Up to 4 months
  To Assessment of Antioxidant Status: TAS (Total Anti-oxydative Status) Levels in Plasma Will Be Measured in Either Waterpipe Smokers or Control Group.
Plasma PON (Paraoxonase) Measurement. | Up to 4 months
  To Assessment of Antioxidant Status: PON Levels in Plasma Will Be Measured in Either Waterpipe Smokers or Control Group.
Plasma sPON (Stimulated Paraoxonase) Measurement. | Up to 4 months
  To Assessment of Antioxidant Status: sPON Levels in Plasma Will Be Measured in Either Waterpipe Smokers or Control Group.
Plasma ARES (Arylesterase) Measurement. | Up to 4 months
  To Assessment of Arylesterase Activity: ARES Levels in Plasma Will Be Measured in Either Waterpipe Smokers or Control Group.

CONTACTS AND LOCATIONS:
Overall Officials: Ozcan Erel, Prof. M.D., Study Director — Ankara Yildirim Beyazit University, Medical School, Director of Biochemistry Department, Ankara, Turkey

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mokdad AH, Warren CW. As if cigarettes were not enough, here comes narghile. A commentary on an article by Yunis et al. in IJPH 52/4. Int J Public Health. 2007;52(5):263-4. doi: 10.1007/s00038-007-0221-6. No abstract available. PMID 18030938
- [Result] Maziak W. The global epidemic of waterpipe smoking. Addict Behav. 2011 Jan-Feb;36(1-2):1-5. doi: 10.1016/j.addbeh.2010.08.030. Epub 2010 Oct 8. PMID 20888700
- [Result] Maziak W, Ward KD, Afifi Soweid RA, Eissenberg T. Tobacco smoking using a waterpipe: a re-emerging strain in a global epidemic. Tob Control. 2004 Dec;13(4):327-33. doi: 10.1136/tc.2004.008169. PMID 15564614
- [Result] Dugas E, Tremblay M, Low NC, Cournoyer D, O'Loughlin J. Water-pipe smoking among North American youths. Pediatrics. 2010 Jun;125(6):1184-9. doi: 10.1542/peds.2009-2335. Epub 2010 May 10. PMID 20457679
- [Result] Shafagoj YA, Mohammed FI. Levels of maximum end-expiratory carbon monoxide and certain cardiovascular parameters following hubble-bubble smoking. Saudi Med J. 2002 Aug;23(8):953-8. PMID 12235470